CLINICAL TRIAL: NCT02038504
Title: a Prospective Study to Investigate the Role of Enteral Nutrition in Nonthyroidal Illness Syndrome Among Fistula Patients
Brief Title: Investigating the Role of EN in NTIS Among Fistula Patients
Acronym: EN;NTIS
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, VIce-president of General Surgery, Jinling Hospital, Professor of Medical School of Nanjing University, Jinling Hospital, China
Other Study IDs: NTIS-EN-1; 81270478 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2014-01-10; First posted 2014-01-16 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Gastrointestinal Fistula
Keywords: gastrointestinal fistula; enteral nutrition; thyroid function
MeSH Terms: conditions — Digestive System Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- gastrointestinal fistula

SUMMARY:
The purpose of this study is to investigate whether enteral nutrition are effective in the treatment of nonthyroidal illness syndrome among fistula patients.

DETAILED DESCRIPTION:
Nonthyroidal illness syndrome (NTIS) is a common alterations in thyroid function observed in about 70% of hospitalized patients, with or without acute systemic illnesses. Mechanisms in the pathogenesis of NTIS are not yet well understood. Our previous study demonstrated that NTIS occurred frequently with a prevalence of 57.5% in gastrointestinal fistulas patients. In recent study, it has been shown that early enteral nutrition decreases the duration of hospitalization and mortality in the burn population, indicating a potential role of enteral nutrition in NTIS.In addition, the management of fistula patients requires bundle therapy including Nutrition therapy, especially enteral nutrition.The purpose of this study is to investigate whether enteral nutrition are effective in the treatment of nonthyroidal illness syndrome among fistula patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastrointestinal fistula
* Clinical diagnosis of nonthyroidal illness syndrome
* Using enteral nutrition for fistula management

Exclusion Criteria:

* patients who were prescribed drug which may affect thyroid function before or in our study
* patients who were diagnosed as primary thyroid disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of general surgery in Jinling hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Thyroid function | Changes of thyroid function from baseline at 1 week,2 week, 3 week and 4 week after enrolled.
  Thyroid function assessment includes level of free triiodothyronine,total triiodothyronine,free thyroxin,total thyroxin,thyroid stimulating hormone,thyroid stimulating hormone index,and standard thyroid stimulating hormone index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Jinling Hospital, Nanjing, Jiangsu, China